CLINICAL TRIAL: NCT01447212
Title: SALOME: Multi-Centre, Double Blind Randomized Controlled Trial Comparing The Effectiveness Of Diacetylmorphine Vs. Hydromorphone For The Treatment Of Long-Term Injection Opioid Users Who Do Not Benefit From Available Therapies
Brief Title: Study to Assess Longer-term Opioid Medication Effectiveness (SALOME)
Acronym: SALOME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Providence Healthcare (Other); Innerchange Charitable Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H09-01455
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Opioid Dependence; Heroin Dependence
Keywords: Opioid Dependence; Long-term Opioid Injectors; Opioid Substitution Treatment; Hydromorphone; Diamorphine; Diacetylmorphine
MeSH Terms: conditions — Opioid-Related Disorders; Heroin Dependence | interventions — Hydromorphone; Injections; Heroin; Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydromorphone (Experimental): Phase I: Injectable Hydromorphone is received for 6 months of the study. Phase II: At 6 months, participants are randomized to either: 1) stay on injectable hydromorphone; or 2) switch to oral hydromorphone, for another six months.
  Interventions: Drug: Hydromorphone, Injectable; Drug: Hydromorphone, liquid oral
- Diacetylmorphine (Active Comparator): Phase I: Injectable Diacetylmorphine is received for 6 months of the study. Phase II: At 6 months, participants are randomized to either: 1) stay on injectable Diacetylmorphine; or 2) switch to oral Diacetylmorphine, for another six months.
  Interventions: Drug: Diacetylmorphine, injectable; Drug: Diacetylmorphine, liquid oral

INTERVENTIONS:
Drug: Hydromorphone, Injectable — Phase I: 3x daily, up to 500mg per day, for 6 months. Phase II: At 6 months, participants are randomized to either: 1) stay on injectable hydromorphone; 2) switch to oral hydromorphone, for another 6 months.
  Arms: Hydromorphone
Drug: Diacetylmorphine, injectable — Phase I: 3x daily, up to 1,000mg per day, for 6 months. Phase II: At 6 months, participants are randomized to either: 1) stay on injectable diacetylmorphine; 2) switch to oral diacetylmorphine, for another 6 months.
  Arms: Diacetylmorphine
Drug: Hydromorphone, liquid oral — Study Phase II: After 6 months of receiving Hydromorphone injectable , participants will be randomized to stay on injectable hydromorphone or switch to oral hydromorphone, for another six months. Oral = experimental; injectable = active comparator
  Arms: Hydromorphone
Drug: Diacetylmorphine, liquid oral — Study Phase II: After 6 months of receiving Diacetylmorphine injectable, participants will be randomized to stay on injectable Diacetylmorphine or switch to oral Diacetylmorphine, for another six months. Oral = experimental; injectable = active comparator
  Arms: Diacetylmorphine

SUMMARY:
The purpose of this study, SALOME, is to determine if 1) the closely supervised provision of injectable, hydromorphone (HDM; trade name Dilaudid™) is as effective as injectable diacetylmorphine (DAM; heroin) in the treatment of chronic, multi-morbid opioid-dependent individuals who have not benefited sufficiently from conventional treatments, and if a switch to the oral equivalent of hydromorphone and diacetylmorphine is as effective as the injection form. The availability of an effective, licensed opioid medication such as hydromorphone, for substitution treatment of chronic, multi-morbid treatment-refractory opioid-dependent individuals, would be of immense impact locally and internationally. It could help to establish alternative treatment options where for non-medical reasons Heroin Assisted Treatment would not be acceptable. Thus, one result could be the expansion of treatment options for the most difficult to treat heroin dependent persons. This would also be an important step for secondary prevention of HIV and Hepatitis C as well as a better integration of those patients in other medical treatments. Switching from intravenous to oral application would also reduce a lot of potential risk factors (like overdose, seizures, infections, etc) and side effects associated with the injection route. Additionally it could make these treatments more feasible in normal treatment settings, like existing methadone services.

DETAILED DESCRIPTION:
SALOME is two-stage single centre (Vancouver) phase III, randomized, double blind controlled trial involving a total of 202 individuals with chronic opioid-dependence who are not benefiting currently from conventional therapies.

Objectives:

The general objectives of this study are to determine whether 1) the closely supervised provision of injectable, hydromorphone is as effective as injectable diacetylmorphine in recruiting, retaining, and benefiting chronic, multi-morbid opioid-dependent individuals who have not benefited sufficient from conventional treatments, and 2) if the switch to the oral equivalent of hydromorphone and diacetylmorphine after six-months is as effective as the injection form.

Secondary outcomes will be evaluated looking at the benefits for the drug users and society of each form of treatment including health status, treatment retention, use of additional methadone, cocaine use and criminal involvement.

Randomization and Treatment Arms:

Stage I: Half of the 202 participants will be randomized to receive injectable diacetylmorphine, and the other half will receive injectable hydromorphone. Stage I will involve 6-months of treatment and the primary outcome will be change in illicit heroin use in the prior 30 days at 6 months.

Stage II: All volunteers retained in injection treatment at the end of Stage I will be eligible to enter Stage II Half the participants will then be randomized to continue injection treatment exactly as in Stage I on a blinded basis while the other half will switch to the oral equivalent of the same medication (diacetylmorphine or hydromorphone). Stage II will involve 6-months of treatment and the primary outcome will be illicit heroin use in the prior 30 days at 6 months after randomization into Stage II.

Individuals completing Stage I will be eligible for Stage II provided they are still receiving injection medication at the treatment clinic. Participants will be excluded from Stage II if they meet any of the exclusion criteria above which may have changed since entry into Stage I. Patients who switch completely to other treatments or abstinence during Stage I will not be randomized to Stage II.

Given that at the present time DAM is not a licensed drug in Canada and HDM for substitution treatment can only be provided as a drug under investigation, at the end of the second study phase patients cannot longer receive these medications. Thus, study treatments will be provided for 12 months followed by a period of up to 1-month during which participants still being treated with DAM or HDM will be tapered and transitioned to conventional therapies such as methadone. From the end of phase two and transitioning period (12 to 13 months) to the next follow-up evaluation (18 month) participants might be receiving Methadone Maintenance Therapy (MMT), engaged in other addiction treatment, abstinent or untreated, using illicit opioids. The 6 and 12-month study visit at which the primary outcome measures will be assessed will be conducted before any tapering or transition began.

Outcomes and follow-up:

Patients will have research assessments performed during the pre-randomization period, at baseline, and at 3, 6, 9, 12, 18 and 24 months following initial randomization The primary outcome measure (POM) for both Stages I and II will be change in illicit heroin use defined as the number of days of illicit ("street") heroin in the prior 30 days of each endpoint (6 months-Stage I, 12 months-Stage II) by means of self report.

Secondary outcome measures will include health status, safety of the study treatments, treatment retention, use of additional methadone, cocaine use, urinalysis, criminal involvement, gender, ethnicity and victimization, health economics and quality of life and an evaluation of the study blinding.

All self-reported outcomes data collection with the study participants will occur in a face-to-face, fully confidential interview setting at the research centre. The interviews will be conducted by trained field research interviewers, who are not part of the clinical treatment team, using standardized instruments. These include: Baseline and follow-up European version of the Addiction Severity Index (EuropASI); EQ-5D (EuroQoL) Opioid Treatment Index (OTI); SCLR-90; WHO Disability Assessment Schedule II (WHO-DAS II); Maudsley Addiction Profile (MAP); Fagerstrom; Health Utilities Index (HUI) as well as Baseline and Follow-up Socio-Demographic questionnaires. The study blinding will be evaluated by a blinding evaluation instrument which follows best practices and current recommendations for evaluating blinding in randomized controlled trials.

ELIGIBILITY:
General Inclusion Criteria:

* Regular use of opioids for five years
* Injecting opioids in the past year
* Two attempts at treatment including one methadone (or other substitution)
* Must be a legal adult
* Struggling with drug related problems

General Exclusion Criteria:

* Pregnancy upon study entry
* Diagnosis of severe medical or psychiatric conditions contra-indicated for diacetylmorphine or hydromorphone treatment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2011-12; Primary Completion 2014-06 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in days of illicit heroin use from baseline. | baseline and 6 months
  Use of illicit heroin at a time point is defined as the number of days of illicit ("street") heroin in the prior 30 days of the 6 month treatment period by means of self report.

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia Oveido-Joekes, Ph.D., Principal Investigator — University of British Columbia; Michael R Krausz, M.D., Principal Investigator — University of British Columbia
Locations (1):
- SALOME Research Office, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Oviedo-Joekes E, Brissette S, Marsh DC, Lauzon P, Guh D, Anis A, Schechter MT. Diacetylmorphine versus methadone for the treatment of opioid addiction. N Engl J Med. 2009 Aug 20;361(8):777-86. doi: 10.1056/NEJMoa0810635. PMID 19692689
- [Background] Oviedo-Joekes E, Guh D, Brissette S, Marsh DC, Nosyk B, Krausz M, Anis A, Schechter MT. Double-blind injectable hydromorphone versus diacetylmorphine for the treatment of opioid dependence: a pilot study. J Subst Abuse Treat. 2010 Jun;38(4):408-11. doi: 10.1016/j.jsat.2010.03.003. Epub 2010 Mar 31. PMID 20359843
- [Derived] Palis H, Marchand K, Guh D, Brissette S, Lock K, MacDonald S, Harrison S, Anis AH, Krausz M, Marsh DC, Schechter MT, Oviedo-Joekes E. Men's and women's response to treatment and perceptions of outcomes in a randomized controlled trial of injectable opioid assisted treatment for severe opioid use disorder. Subst Abuse Treat Prev Policy. 2017 May 19;12(1):25. doi: 10.1186/s13011-017-0110-9. PMID 28526048
- [Derived] Oviedo-Joekes E, Guh D, Brissette S, Marchand K, MacDonald S, Lock K, Harrison S, Janmohamed A, Anis AH, Krausz M, Marsh DC, Schechter MT. Hydromorphone Compared With Diacetylmorphine for Long-term Opioid Dependence: A Randomized Clinical Trial. JAMA Psychiatry. 2016 May 1;73(5):447-55. doi: 10.1001/jamapsychiatry.2016.0109. PMID 27049826
- [Derived] Oviedo-Joekes E, Marchand K, Lock K, MacDonald S, Guh D, Schechter MT. The SALOME study: recruitment experiences in a clinical trial offering injectable diacetylmorphine and hydromorphone for opioid dependency. Subst Abuse Treat Prev Policy. 2015 Jan 26;10:3. doi: 10.1186/1747-597X-10-3. PMID 25619263